CLINICAL TRIAL: NCT03384212
Title: CBA Versus FBA Conditioning Followed by Allogeneic HSCT in Treatment of High Risk and Refractory AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Changhai Hospital (Other); Xiangya Hospital of Central South University (Other); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Chengdu PLA General Hospital (Other); Tang-Du Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Chun Wang, director, department of hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-22
Record Dates: First submitted 2017-11-05; First posted 2017-12-27 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: High Risk Acute Myeloid Leukemia; Allogeneic Hematopoeitic Stem Cell Transplantation
Keywords: cladribine; fludarabine; relapse
MeSH Terms: conditions — Recurrence | interventions — Cladribine; fludarabine; Busulfan; Cytarabine

STUDY DESIGN:
Intervention Model Description: open labled randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBA group (Experimental): CBA as HSCT conditioning:
  cladribine 5mg/m2 day -6 to day -2 busulfan(iv) 3.2mg/kg day-6 to day -3 cytarabine 2g/m2 day-6 to day -2
  Interventions: Drug: Cladribine; Drug: Busulfan; Drug: Cytarabine
- FBA group (Active Comparator): FBA as HSCT conditioning:
  fludarabine 30mg/m2 day -6 to day -2 busulfan(iv) 3.2mg/kg day-6 to day -3 cytarabine 2g/m2 day-6 to day -2
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Cytarabine

INTERVENTIONS:
Drug: Cladribine
  Other Names: chlorodeoxyadenosine
  Arms: CBA group
Drug: Fludarabine
  Arms: FBA group
Drug: Busulfan
  Other Names: busulphan
Drug: Cytarabine
  Other Names: cytosine arabinoside

SUMMARY:
Aim: To evaluated if cladribine based conditioning (CBA) could decrease relapse after HLA matched HSCT in high risk and refractory AML patients as compared with fludarabine based conditioning regimen(FBA).

Study design: open-labed, prospective, multicenter, randomized control study Number of subjects: 60 each group

Treatment:

CBA group: CBA as HSCT conditioning which including cladribine 5mg/m2 day -6 to day -2 , busulfan(iv) 3.2mg/kg day-6 to day -3 and cytarabine 2g/m2 day-6 to day -2.

FBA group: FBA as HSCT conditioning which including fludarabine 30mg/m2 day -6 to day -2, busulfan(iv) 3.2mg/kg day-6 to day -3 and cytarabine 2g/m2 day-6 to day -2.

DETAILED DESCRIPTION:
Relapse is still the main reason of death for patients with acute myeloid leukemia (AML) undergoing allogeneic hematopoietic stem cell transplantation (HSCT), especially for those with high risk and refractory disease. Cladribine and fludarabine are both purine analogs used in treatment of AML. Two studies by the Polish Adult Leukemia Group (PALG) demonstrated that the addition of cladribine to DA (DAC) was associated with an increased complete remission (CR) rate and prolonged overall survival (OS) in the general AML population, with the most prominent effect in patients with unfavorable cytogenetics. Therefore we presume cladribine may more effective in eliminating leukemic cells so that reduce relapse after HSCT.

Eligible patients in this study should between 18 to 60 years old with confirmed AML and fulfilled at least one criteria defining high risk or refractory disease.Patients must have HLA 9/10 or 10/10 matched sibling or unrelated donor. Patients will be excluded if they present any contraindication for HSCT, including respiratory failure, heart failure, liver or kidney function failure et al.

To evaluate if cladribine based conditioning (CBA) could decrease relapse after HLA matched HSCT in high risk and refractory AML patients as compared with fludarabine based conditioning regimen(FBA), 120 eligible patients will be randomized to two groups, the CBA group and the FBA group. Patients in the CBA group receive conditioning including cladribine 5mg/m2 day -6 to day -2 , busulfan(iv) 3.2mg/kg day-6 to day -3 and cytarabine 2g/m2 day-6 to day -2. While patients in the FBA group receive conditioning including fludarabine 30mg/m2 day -6 to day -2 , busulfan(iv) 3.2mg/kg day-6 to day -3 and cytarabine 2g/m2 day-6 to day -2. Graft versus host disease(GVHD) prophylactic regimen include cyclosporine A and short term MTX, ATG 6mg/kg is additionally administered to patients with unrelated donors.

Patients will be followed up for 2 years and the primary end point is the cumulative relapse rate at 2 years. The second end points of the study include the overall survival, disease free survival and non-relapse mortality at 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML confirmed by bone marrow cell morphology, immunology, cytogenetics and molecular biology (MICM). Blast crisis of chronic myeloid leukemia (CML) and AML transferred from myelodysplastic syndrome(MDS) or other diseases are also included.
2. AML with high risk cytogenetic abnormals, such as FLT3- ITD, et al.
3. Patients fulfilled at least one of the following criteria defining refractory AML:(1) primary induction failure (PIF) after 2 or more cycles of chemotherapy; (2) first early relapse after a remission duration of fewer than 12 months and refractory to salvage combination chemotherapy; (3) second or subsequent relapse .
4. Have HLA 9/10 or 10/10 matched siblings or unrelated donor，the donor must match the health conditions of hematopoietic stem cell donation (criteria of China Marrow Donor Program) and be willing to donate.
5. Performance status score no more than 2 (ECOG criteria).
6. Adequate organ function as defined by the following criteria:ALT, AST and total serum bilirubin <2×ULN (upper limit of normal), Serum creatinine and BUN <1.25×ULN.
7. Adequate cardiac function without acute myocardial infarction, arrhythmia or atrioventricular block, heart failure, active rheumatic heart disease and cardiac dilatation.
8. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
9. Willingness and ability to comly with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Presence of any condition inappropriate for HSCT.
2. Presence of any fatal disease, including respiratory failure, heart failure, liver or kidney function failure et al.
3. Have no suitable donor.
4. Pregnancy or breast feeding.
5. Current treatment on another clinical trail.
6. Any other condition the investigator judged the patient inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
cumulative relapse rate at 2 year | 2 years
  The percentage of all patients who are relapsed within 2 years after allogeneic HSCT.

SECONDARY OUTCOMES:
overall survival at 2 year | 2 years
  The percentage of all patients who are still alive 2 years after allogeneic HSCT.
disease free survival at 2year | 2 years
  The percentage of all patients who are leukemia free 2 years after allogeneic HSCT.
non-relapse mortality at 2year | 2 years
  The percentage of patients who are dead of all reasons except relapse.
non-relapse mortality at 100days | 100 days
  The percentage of patients who are dead of all reasons except relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, M.D.,Ph. D., Study Chair — Shanghai General Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Shanghai general hospital, Shanghai Jiaotong university school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holowiecki J, Grosicki S, Robak T, Kyrcz-Krzemien S, Giebel S, Hellmann A, Skotnicki A, Jedrzejczak WW, Konopka L, Kuliczkowski K, Zdziarska B, Dmoszynska A, Marianska B, Pluta A, Zawilska K, Komarnicki M, Kloczko J, Sulek K, Haus O, Stella-Holowiecka B, Baran W, Jakubas B, Paluszewska M, Wierzbowska A, Kielbinski M, Jagoda K; Polish Adult Leukemia Group (PALG). Addition of cladribine to daunorubicin and cytarabine increases complete remission rate after a single course of induction treatment in acute myeloid leukemia. Multicenter, phase III study. Leukemia. 2004 May;18(5):989-97. doi: 10.1038/sj.leu.2403336. PMID 14999298
- [Background] Holowiecki J, Grosicki S, Giebel S, Robak T, Kyrcz-Krzemien S, Kuliczkowski K, Skotnicki AB, Hellmann A, Sulek K, Dmoszynska A, Kloczko J, Jedrzejczak WW, Zdziarska B, Warzocha K, Zawilska K, Komarnicki M, Kielbinski M, Piatkowska-Jakubas B, Wierzbowska A, Wach M, Haus O. Cladribine, but not fludarabine, added to daunorubicin and cytarabine during induction prolongs survival of patients with acute myeloid leukemia: a multicenter, randomized phase III study. J Clin Oncol. 2012 Jul 10;30(20):2441-8. doi: 10.1200/JCO.2011.37.1286. Epub 2012 Apr 16. PMID 22508825